CLINICAL TRIAL: NCT00089024
Title: A Phase II Study Of Neo-Adjuvant Chemotherapy And Radiation In Patients With Locally Advanced Pancreatic Cancer
Brief Title: Combination Chemotherapy, and Radiation Therapy in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0035-04-FB; P30CA036727 (NIH)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Fluorouracil; Gemcitabine; Leucovorin; Folic Acid Antagonists; Oxaliplatin; Drug Therapy; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental): see interventions
  Interventions: Drug: fluorouracil; Drug: gemcitabine hydrochloride; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: adjuvant therapy; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy

INTERVENTIONS:
Drug: fluorouracil — 2700 mg/m5 IV over 24 hr after gemcitabine weeks 1 & 2; Repeat one 3-week cycle starting day 22
  Other Names: Tolak, Fluoroplex, Carac
Drug: gemcitabine hydrochloride — 750 (females) or 900 (males) mg/m5 IV over 30 min (day 2)weeks 1 & 2; Repeat one 3-week cycle starting day 22
  Other Names: Gemzar
Drug: leucovorin calcium — 20 mg/m5 PO (day 1) and 20 mg/m5 IV (day 2) weeks 1 and 2; Repeat one 3-week cycle starting day 22
  Other Names: folic acid analog
Drug: oxaliplatin — 48 mg/m5 IV over 2 hr weeks 1, 2, 4, and 5
  Other Names: chemotherapy
Procedure: adjuvant therapy — Patients who have undergone surgical resection, after post-operative recovery, will receive two additional cycles of gemcitabine/5-FU/leucovorin. Patients will then be followed at 3 month intervals with a history and physical exam, CT scan of the chest/abdomen/pelvis, and tumor markers.
  If surgical resection is not possible, patients with stable or responsive disease will resume gemcitabine/5-FU/leucovorin and continue on it indefinitely until disease progression provided the patient tolerates it and wishes to remain on therapy.
Procedure: conventional surgery — Restaging with repeat imaging studies will be performed four weeks after completion of the chemo-radiation. If no contraindication for surgical resection is identified, resection will be performed six to eight weeks after completing chemoradiation. At the time of surgical resection, an extensive examination of the abdomen will be performed to exclude the presence of metastatic disease. All operations will be performed with curative intent with resection of all gross tumor (ie R0 [negative margins] or R1 [positive microscopic margins]). Resection of adjacent involved organs or vascular structures will be performed as clinically indicated.
Procedure: neoadjuvant therapy — Eligible patients will receive an initial two cycles of chemotherapy with gemcitabine 750 (females) or 900 (males) mg/m5 over 30 minutes followed by a 24-hour infusion of fluorouracil 2700 mg/m5 on days 2 and 9 of a 21-day cycle . Calcium leucovorin 20 mg/m5 will be given orally on days 1 and 8 and by IV push on days 2 and 9 prior to the 5-FU. A window of -2 up to +7 days will be allowed to start planned cycles of therapy provided all other criteria to restart the new cycle has been met. Patients will require a central venous catheter (Port, Hickman or Groshong catheter) for the administration of 5-FU.
Radiation: radiation therapy — A re-staging CT scan, which will be obtained as part of the radiation simulation, will be used to assess any possible response to the initial two cycles of chemotherapy. Unless the patient has developed evidence of metastatic disease, chemoradiation will proceed. Patients who required no treatment delays will commence chemoradiation on day 42. If a one-week delay is needed before cycle 2 of neo-adjuvant chemotherapy can be delivered, the patient will begin chemoradiation on day 49 provided treatment-related toxicity has resolved. If cycle 2 could not be given (2 or more week delay for resolution of treatment-related toxicity), then chemoradiation will begin once toxicity has resolved (may be earlier than day 42).

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving combination chemotherapy with radiation therapy before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with radiation therapy works in treating patients who may undergo surgery for locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor and clinical benefit response to neoadjuvant chemoradiotherapy comprising gemcitabine, fluorouracil, leucovorin calcium, and oxaliplatin in patients with potentially resectable locally advanced adenocarcinoma of the pancreas.
* Determine the toxic effects of this regimen in these patients.
* Determine the achieved steady-state plasma levels of gemcitabine and fluorouracil in these patients and correlate these plasma levels with clinical toxicity associated with this regimen.
* Determine the potential importance of polymorphic variations in genomic DNA of pertinent genes (whose protein products are targets of the antineoplastic drugs used in this study) on response to and toxicity of this regimen in these patients.
* Determine the gene expression profiles of primary and metastatic pancreatic tumors before and after treatment with this regimen.

OUTLINE:

* Neoadjuvant chemotherapy: Patients receive gemcitabine IV over 30 minutes and fluorouracil IV continuously over 24 hours on days 2 and 9, and leucovorin calcium orally on days 1 and 8 and IV on days 2 and 9. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
* Neoadjuvant chemoradiotherapy: Beginning on day 42, patients undergo chemoradiotherapy comprising oxaliplatin IV over 2 hours on days 42, 49, 56, 63, 70, and 77 and fluorouracil IV continuously on days 42-78 with external beam radiotherapy.
* Surgery: Patients undergo surgical resection 42-56 days after completion of chemoradiotherapy.
* Adjuvant chemotherapy: After post-operative recovery, patients receive 2 additional courses of gemcitabine, fluorouracil, and leucovorin calcium. If surgical resection is not possible, patients with stable or responsive disease resume gemcitabine, fluorouracil, and leucovorin calcium indefinitely in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the pancreas

  o Locally advanced disease
* Potentially resectable disease
* 19 years of age and over
* Karnofsky 60-100%
* Absolute granulocyte count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 2.0 mg/dL (in the absence of biliary obstruction)

  * If biliary obstruction is present, patients must undergo biliary decompression
  * Bilirubin ≤ 3.0 mg/dL after biliary drainage has been established
* Creatinine ≤ 1.6 mg/dL

Exclusion Criteria:

* No early stage resectable disease
* No concurrent non-steroidal anti-inflammatory medication
* No evidence of distant metastases to the liver or peritoneal area according to imaging studies and laparoscopic staging
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No serious uncontrolled cardiac arrhythmia
* Not pregnant or nursing
* No uncontrolled illness
* No active or ongoing infection requiring IV antibiotics
* No marked intolerance to 5-fluoropyrimidines (i.e., fluorouracil, floxuridine, capecitabine, or fluorocytosine)
* No allergy to sulfonamides, aspirin, or non-steroidal anti-inflammatory drugs
* No allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with study chemotherapy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated noninvasive carcinoma
* No prior chemotherapy for pancreatic cancer
* No prior abdominal radiotherapy

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-02-25 (Actual); Primary Completion 2010-01-22 (Actual); Study Completion 2014-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Grem, MD, Study Chair — University of Nebraska
Locations (1):
- Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: neoadjuvant regimen involving gemcitabine, infusional 5-fluorouracil (5-FU), oxaliplatin and radiation therapy (RT) in patients with potentially resectable locally advanced pancreatic adenocarcinoma.
  Induction chemotherapy (CT) consisted of two 3-week cycles of weekly gemcitabine with 24-hour continuous infusion of 5 FU for 2 of 3 weeks. Chemoradiation (CRT) consisted of RT of 50.4 Gy in 28 fractions or 50 Gy in 25 fractions and weekly oxaliplatin with 24-hour continuous infusion of 5 FU throughout RT. The first 7 patients also received celecoxib 200 mg BID throughout induction CT and CRT.
Period: Overall Study
Arm/Group | Treatment
Started | 29
Treated Subjects | 29
Completed | 24
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] — Analysis is of the 29 subjects that consented and initiated treatment.
  years | 60 [49 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 28
  Hispanic | 1

OUTCOME MEASURES:

1. Primary Outcome: Surgical Exploration
Description: Patients who completed chemotherapy & chemo-radiation had restaging imaging studies 4 weeks after completion of chemo-radiation. If there were no contraindications for surgical resection, surgical exploration was performed 6-8 weeks after completing chemo-radiation
Time Frame: After 6 weeks of chemotherapy and then after 4 weeks of chemo-radiation.
Population: Only 19 participants under went surgical exploration.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Eligible patients will receive an initial two cycles of chemotherapy with: gemcitabine 750 (females) or 900 (males) mg/m5 over 30 minutes followed by a 24-hour infusion of fluorouracil 2700 mg/m5 on days 2 and 9 of a 21-day cycle . Calcium leucovorin 20 mg/m5 will be given orally on days 1 and 8 and by IV push on days 2 and 9 prior to the 5-FU.
  Radiation therapy: Patients who required no treatment delays will commence chemoradiation on day 42.
  Restaging with repeat imaging studies will be performed four weeks after completion of the chemo-radiation. Resection will be performed six to eight weeks after completing chemoradiation.
  Patients who have undergone surgical resection, after post-operative recovery, will receive two additional cycles of gemcitabine/5-FU/leucovorin. If surgical resection is not possible, patients with stable or responsive disease will resume gemcitabine/5-FU/leucovorin and continue on it indefinitely until disease progression
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants
  unresectable disease | 4
  intra-abdominal metastasis | 6
  resection of the primary tumor | 9

2. Primary Outcome: Number of Participants Experiencing Grade 3-4 Toxicity While Receiving the Study Treatment
Description: Toxicity event collected during Induction chemotherapy (CT) - two 3-week cycles, Concurrent CT and Radiation Therapy (CRT) (approximately 5.5 weeks), post CRT (4 weeks after the end of CRT), 2-3 months post CRT (8-12 weeks after the end of CRT)
Time Frame: From time of first dose until 30 days following final treatment, approximately 24 weeks
Population: A total of 29 patients started induction CT. Two patients dropped out because of progressive disease (PD) and 1 died from pulmonary embolus. 27 patients continued with CRT 24 (89%) received the full radiation dose. Of 24, 5 went off study prior to surgical exploration, for remaining 19 with surgical exploration.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 29
Participants
  Induction CT, grade 3 | 4
  Induction CT, grade 4 | 5
  CRT, grade 3: number analyzed (Participants) | 27
  CRT, grade 3 | 11
  CRT, grade 4: number analyzed (Participants) | 27
  CRT, grade 4 | 0
  Within 1 mo. post CRT, grade 3: number analyzed (Participants) | 27
  Within 1 mo. post CRT, grade 3 | 12
  Within 1 mo. post CRT, grade 4: number analyzed (Participants) | 27
  Within 1 mo. post CRT, grade 4 | 1
  2-3 mos. post CRT, grade 3: number analyzed (Participants) | 19
  2-3 mos. post CRT, grade 3 | 9
  2-3 mos. post CRT, grade 4: number analyzed (Participants) | 19
  2-3 mos. post CRT, grade 4 | 0

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events from the time of first treatment until they 30 days after last day of study treatment. (approximately 24 weeks)
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 7/29
Serious Adverse Events (participants affected / at risk) | 25/29
Other Adverse Events (participants affected / at risk) | 27/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=29)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — bloody stool
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — liver abscess
Sepsis (Infections and infestations) | 4 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) — gastrointestinal bleed
Myocardial infarction (Cardiac disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) — thrombus
Investigations - Other, specify (Investigations) | 2 (2) — hemoglobin
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) — Failure to thrive
Investigations - Other, specify (Investigations) | 1 (1) — tachycardia
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) — pulmonary emboli
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — septic shock
Ascites (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) — hemolytanemia
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — chyle leak
Investigations - Other, specify (Investigations) | 1 (1) — bilirubin
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) — platelets
Gastrointestsinal disorders - other, specify (Gastrointestinal disorders) | 1 (1) — Perforation of gastrojejunostomy site
Gastrointestinal disorders- Other, specify (Gastrointestinal disorders) | 1 (1) — Enterocutaneous fistula
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — gastroenteritis
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — biliary obstruction
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) — epigastric pain
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — presyncopal episode
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) — cholangitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=29)
Thromboembolic event (Vascular disorders) | 8 (9)
Fatigue (General disorders) | 7 (8)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4 (4) — Failure to thrive
Nausea (Gastrointestinal disorders) | 5 (5)
Hemoglobin (Investigations) | 8 (9)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 6 (27) — Neutropenia
Hyponatremia (Metabolism and nutrition disorders) | 10 (15)
Urinary tract infection (Infections and infestations) | 2 (2)
Investigations - Other, specify (Investigations) | 5 (5) — GGT
Hypokalemia (Metabolism and nutrition disorders) | 12 (22)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (4) — weakness
Investigations - Other, specify (Investigations) | 5 (5) — Bilirubin
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Investigations - Other, specify (Investigations) | 2 (2) — alanine aminotransferase
Abdominal Pain (Gastrointestinal disorders) | 3 (6)
Renal and urinary disorders - Other, specity (Renal and urinary disorders) | 2 (2) — acute renal failure
Investigations - Other, specify (Investigations) | 2 (2) — alkaline phosphatase
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Investigations - Other, specify (Investigations) | 2 (2) — aspartate aminotransferase
Investigations - Other, specify (Investigations) | 2 (2) — bacteremia
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (7)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (12) — leukopenia
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) — Pulmonary embolism
Sepsis (Infections and infestations) | 3 (3)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (4) — thrombocytopenia
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (Investigations) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes